CLINICAL TRIAL: NCT04164550
Title: Postoperative Complications, Nasal Function, and Quality of Life Following Interpolated Flap Repair for Post-Mohs Surgical Defects of the Nose: a Multi-center Prospective Observational Cohort Study
Brief Title: Interpolated Flap Study
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Oregon Health and Science University (Other); Stanford University (Other); University of Minnesota (Other); University of Missouri-Columbia (Other); University of Vermont (Other); University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 829285
Record Dates: First submitted 2019-11-05; First posted 2019-11-15 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Skin Cancer, Non-Melanoma; Skin Cancer Melanoma; Mohs Micrographic Surgery
MeSH Terms: conditions — Skin Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary purpose of this study is to address the limited knowledge regarding patient well- being and nasal function after interpolated flap repair of post-Mohs surgical defects on the nose. Improved understanding of the patient experience will allow providers to better counsel their patients pre-operatively and potentially identify patients who may benefit from additional interventions.

DETAILED DESCRIPTION:
This project is a multi-center prospective cohort study evaluating postoperative complication rates, quality of life outcomes, and nasal function after interpolated flap repair of post-Mohs surgical defects of the nose. Our primary outcome is the incidence of short-term complications(within 4 weeks of surgery) defined by the American College of Mohs Surgery as: death, bleeding requiring additional intervention, functional loss attributable to surgery, hospitalization for an operative complication, and surgical site infection. Secondary outcomes will include incidence of flap necrosis and evaluation of quality of life at 1, 4 and 16 weeks after repair. Quality of life will be investigated using the Skin Cancer Index (SCI)- a skin cancer specific quality of life instrument and the Nasal Appearance and Functional Evaluation Questionnaire (NAFEQ). Previous literature has demonstrated that Mohs surgery in the outpatient setting has a very low complication rate but this literature is generally limited to single-institution studies or studies examining smaller repairs. Furthermore, it has been proven that receiving a skin cancer diagnosis is stressful and patient satisfaction with skin cancer surgery is related to their appearance and scarring or changes in appearance can decrease quality of life. Our study serves to fill the current literature knowledge gaps by examining repair of large defects and looking at both complications and quality of life outcomes. Data collection will begin pre-operatively on patients 18 and older who require an interpolated flap repair of a post-Mohs surgical defect. These patients will then be followed and asked to complete SCI and NAFEQ surveys as well as complication questionnaires at prescribed intervals. All data will be stored via a secure RedCap database.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older who are able to provide informed consent and may require interpolated flap repair of their post-Mohs surgical defect

Exclusion Criteria:

* People who are not adults, not able to give informed consent, or who's wounds are not being repaired by a fellowship trained Mohs surgeon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients age 18 years or greater who are capable of providing informed consent and who may require an interpolated flap repair of their post-Mohs surgical defect will be recruited. If they consent to the study, they will be asked to complete the SCI and NAFEQ preoperatively. Patients who subsequently undergo interpolated flap repair will be followed and will complete subsequent SCI and NAFEQ surveys at one week from the date of the interpolated flap inset, 4 weeks after flap takedown, and 16 weeks after flap takedown. The target enrollment is 180 patients undergoing interpolated flap repair.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Complication rate following Mohs micrographic surgery and flap inset | 30 days
  Short term (30 day) complications are defined by the American College of Mohs Surgery as death, bleeding requiring additional intervention, functional loss attributable to surgery, hospitalization for an operative outcome, and surgical site infection.
Complication rate following flap takedown | 30 says
  Short term (30 day) complications are defined by the American College of Mohs Surgery as death, bleeding requiring additional intervention, functional loss attributable to surgery, hospitalization for an operative outcome, and surgical site infection.

SECONDARY OUTCOMES:
One week after Mohs- Skin Cancer Index Score | 1 week after Mohs micrographic surgery
  Skin Cancer Index is 15-item, disease specific, validated, quality of life instrument with three sub-scales, Emotion, Social, Appearance. A 5-point response format is used for each question where 1 equals "very much" and 5 equals "not at all". Standardized Scores Range from 0-100 with higher scores indicating higher quality of life. Standardized scores are obtained by summing the individual scores and dividing them by the number of items in each sub-scale.
Four weeks after flap takedown- Skin Cancer Index Score | 4 weeks after flap takedown surgery
  Skin Cancer Index is 15-item, disease specific, validated, quality of life instrument with three sub-scales, Emotion, Social, Appearance. A 5-point response format is used for each question where 1 equals "very much" and 5 equals "not at all". Standardized Scores Range from 0-100 with higher scores indicating higher quality of life. Standardized scores are obtained by summing the individual scores and dividing them by the number of items in each sub-scale.
Sixteen weeks after flap takedown- Skin Cancer Index Score | 16 weeks after flap takedown surgery
  Skin Cancer Index is 15-item, disease specific, validated, quality of life instrument with three sub-scales, Emotion, Social, Appearance. A 5-point response format is used for each question where 1 equals "very much" and 5 equals "not at all". Standardized Scores Range from 0-100 with higher scores indicating higher quality of life. Standardized scores are obtained by summing the individual scores and dividing them by the number of items in each sub-scale.
One week after Mohs- Nasal Appearance and Functional Evaluation Questionnaire (NAFEQ) Score | 1 week after Mohs micrographic surgery
  The NAFEQ is a 14-item, validated quality of life instrument with two sections. The first seven items regard nasal function and airway passage, while the following seven questions assess satisfaction with nasal appearance. Responses are rated on a 5-point Likert scale where 1 equals "always" or "very dissatisfied", depending on the question, and 5 equals "never" or "very satisfied". Potential scores range from 7-35 with higher scores indicating greater satisfaction with overall nasal functioning and appearance.
Four weeks after flap takedown- Nasal Appearance and Functional Evaluation Questionnaire (NAFEQ) Score | 4 weeks after flap takedown surgery
  The NAFEQ is a 14-item, validated quality of life instrument with two sections. The first seven items regard nasal function and airway passage, while the following seven questions assess satisfaction with nasal appearance. Responses are rated on a 5-point Likert scale where 1 equals "always" or "very dissatisfied", depending on the question, and 5 equals "never" or "very satisfied". Potential scores range from 7-35 with higher scores indicating greater satisfaction with overall nasal functioning and appearance.
Sixteen weeks after flap takedown- Nasal Appearance and Functional Evaluation Questionnaire (NAFEQ) Score | 16 weeks after flap takedown surgery
  The NAFEQ is a 14-item, validated quality of life instrument with two sections. The first seven items regard nasal function and airway passage, while the following seven questions assess satisfaction with nasal appearance. Responses are rated on a 5-point Likert scale where 1 equals "always" or "very dissatisfied", depending on the question, and 5 equals "never" or "very satisfied". Potential scores range from 7-35 with higher scores indicating greater satisfaction with overall nasal functioning and appearance.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Etzkorn, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided